CLINICAL TRIAL: NCT06382545
Title: Post-instrumentation Pain After Use of the Fanta and M3 Pro Gold Systems: A Randomized Clinical Trial
Brief Title: Post-instrumentation Pain After Use of the Fanta and M3 Pro Gold Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Faten Mohamed Ahmed Ghonimy, Assisstany Professor, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Approval number 36.3.22
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Endodontic Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 participants treated with Fanta (Pepsi gold) (FPG) (Experimental): aged 20 to 50 years
  Interventions: Procedure: Fanta (Pepsi gold) (FPG)
- 20 participants treated with M3-pro+ Gold (assorted) (MPG) rotary files (Experimental): aged 20 to 50 years
  Interventions: Procedure: M3-pro+ Gold (assorted) (MPG)

INTERVENTIONS:
Procedure: Fanta (Pepsi gold) (FPG) — endodontic treatment of posterior teeth with Fanta (Pepsi gold) (FPG)
  Arms: 20 participants treated with Fanta (Pepsi gold) (FPG)
Procedure: M3-pro+ Gold (assorted) (MPG) — endodontic treatment of posterior teeth with M3-pro+ Gold (assorted) (MPG) rotary files.
  Arms: 20 participants treated with M3-pro+ Gold (assorted) (MPG) rotary files

SUMMARY:
Comparing the intensity of post-operative pain following endodontic treatment of posterior teeth with Fanta (Pepsi gold) (FPG) and M3-pro+ Gold (assorted) (MPG) rotary files.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old
* No systemic diseases
* Mandibular first molar
* Asymptomatic tooth
* Normal periapical film
* Restorable teeth
* Periodontal scoring index <2

Exclusion Criteria:

* Age <20 and >50
* Systemic disorders
* Articaine Allergy
* Inability to take paracetamol.
* Pregnancy or Nursing
* Symptomatic pulpitis.
* Pulp necrosis
* PDL is widening.
* Periapical radiolucency
* The sinus tract
* Periapical abscesses.
* Existence of resorption
* Tooth malposition.
* Fixed partial dentures.
* Analgesics intake in the last 12 hours.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
comparing the intensity of post-instrumentation pain | The patients were referred for treatment over a period of 7 months from November 2021-May 2022.
  Participants were asked to assign a Visual Analoge Scale (VAS) score to their reported pain. The existence or absence of pain was classified into four groups: no pain (0), mild pain (1-3), moderate pain (4-6), and severe pain (7-10), following endodontic treatment of posterior teeth with Fanta (Pepsi gold) (FPG) and M3-pro+ Gold (assorted) (MPG) rotary files.

CONTACTS AND LOCATIONS:
Overall Officials: Faten Ghonimy, Study Director — Ahram Canadian University
Locations (1):
- Faculty of Oral and Dental medicine, Ahram Canadian University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes